CLINICAL TRIAL: NCT04391504
Title: Intracardiac Versus Transesophageal Echocardiography for Left Atrial Appendage Occlusion Combined With Radiofrequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruiqin xie (Other)
Responsible Party: Sponsor-Investigator, Ruiqin xie, director of cardiology department, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XieruiqindoctorLAA
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
Keywords: transesophageal echocardiography; intracardiac echocardiography; left atrial appendage closure combined with radiofrequency ablation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: A total of 60 patients with atrial fibrillation were scheduled to receive left atrial appendage occlusion combined with radiofrequency ablation, which were divided into two groups. The operation was performed under the guidance of intracardiac echocardiography and transesophageal echocardiography respectively (allocation ratio 1:1).
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers will participate in the operation to record operative parameters. Other researchers including follow-up personnel and the ultrasonic data analyst are uninformed about the random situation of the patients (patient information is recorded according to the random number.Random numbers corresponding to the random allocation list are stored in the research center. After follow-up of the last patient is completed, the random allocation list is published by the random number designer; and the designer does not participate in the data collection and statistics.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transesophageal echocardiography guidance (Experimental)
  Interventions: Procedure: LAAC combined with radiofrequency ablation group
- intracardiac echocardiography guidance (Experimental)
  Interventions: Procedure: LAAC combined with radiofrequency ablation group

INTERVENTIONS:
Procedure: LAAC combined with radiofrequency ablation group — Each patient received the same group of patients with simple radiofrequency ablation radiofrequency ablation treatment at the same time, the transcatheter occlusion of left atrial appendage opening

SUMMARY:
A total of 60 patients with atrial fibrillation were scheduled to receive left atrial appendage occlusion combined with radiofrequency ablation, which were divided into two groups. The operation was performed under the guidance of intracardiac echocardiography and transesophageal echocardiography respectively (allocation ratio 1:1). During the operation, the total amount of contrast medium injected, the fluoroscopy time and the time from femoral vein puncture to transseptal puncture to closure were recorded in all patients. All patients underwent transesophageal echocardiography before and 3 months after operation, and the results were explained by two experienced ultrasound doctors to measure the presence of left atrial thrombus, residual shunt and device-related thrombus. All patients were examined by transthoracic echocardiography 3 months after operation to evaluate new pericardial effusion, pericardial tamponade, instrument embolization / displacement and so on. The baseline clinical and surgical features and hospitalization outcomes of patients guided by ICE and TEE were recorded and compared. Clinical endpoints include death, new pericardial effusion that does not require pericardiocentesis, tamponade with pericardiocentesis, instrument embolism / displacement, bleeding at the entry site, thromboembolic events (stroke / transient ischemic attack [TIA]), and renal failure requiring dialysis. The purpose of this study was to evaluate the feasibility, safety and effectiveness of intracardiac echocardiographic (ICE)-guided and transesophageal echocardiographic (TEE)-guided left atrial appendage occlusion combined with radiofrequency ablation. And try to analyze whether intracardiac echocardiography can be used as an alternative to transesophageal echocardiography in transcatheter closure of left atrial appendage. The average follow-up time was 1 year.

ELIGIBILITY:
Inclusion Criteria:

sustained AF attack occurred in patients with a duration of more than one year, patients taking class I and class III antiarrhythmic drugs could not prevent AF, patients younger than 80 years old Cha2ds2-vasc score ≥2, not suitable for long-term oral anticoagulant drugs.

Exclusion Criteria:

Patients with a history of atrial thrombosis or valvular heart disease (moderate or severe valve stenosis or severe valve regurgitation), patients undergoing prosthetic heart valve replacement, pregnant women, patients with previous liver and kidney diseases, malignant tumors or blood system diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
injected contrast media as well as fluoroscopy time were recorded | in the procedure
  injected contrast media as well as fluoroscopy time were recorded in all patients
the time from femoral vein puncture to transseptal puncture to closure were recorded | in the procedure
  the time from femoral vein puncture to transseptal puncture to closure were recorded in all patients
residual shunt and DRT after transcatheter closure of left atrial appendage detected | 1-12months
  Transesophageal echocardiography
new pericardial effusion, pericardial tamponade were detected | 1-12months
  Transthoracic echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Liu Q, You L, Yang J, Zhang Y, Wu J, Yin H, Zhang Y, Xie R. Clinical Results and Safety of Intracardiac Echocardiography Guidance for Combined Catheter Ablation and Left Atrial Appendage Occlusion. Rev Cardiovasc Med. 2024 May 27;25(6):192. doi: 10.31083/j.rcm2506192. eCollection 2024 Jun. PMID 39076324